CLINICAL TRIAL: NCT03056625
Title: Efficacy of Vitamin A Fortified Rice in Lactating Thai Women
Acronym: EVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Siwaporn Pinkaew, Principal investigator, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MGR5980155
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Vitamin A Status
Keywords: fortified rice; lactating women; 13C2-retinol isotope dilution; vitamin A liver store

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortified rice (Experimental): Participant will be given vitamin A fortified rice 1 meal/day
  Interventions: Other: Vitamin A fortified rice
- Control (Placebo Comparator): Participant will be given normal rice 1 meal/day
  Interventions: Other: Normal rice

INTERVENTIONS:
Other: Vitamin A fortified rice — Lactating women will receive fortified rice one meal per day on weekdays for a period of 14 weeks.
  Arms: Fortified rice
Other: Normal rice — Lactating women will receive normal rice one meal per day on weekdays for a period of 14 weeks.
  Arms: Control

SUMMARY:
Vitamin A deficiency (VAD) remains a public health problem that occurs in children and women. WHO estimates that 190 million preschool age children (under five years of age) and 19.1 million pregnant women have inadequate concentrations of retinol . VAD may increase risk of morbidity and mortality during childhood, pregnancy and postpartum period . In developing countries, vitamin A status in lactating women is not optimal. Even in the United States, vitamin A status of low income pregnant women is marginal. Therefore, women of reproductive age are at risk of vitamin A depletion which compromises the vitamin A status of breastfed infants. Vitamin A is transferred to milk from both retinol binding protein bound and chylomicron associated vitamin A carriers. Because of teratogenicity of vitamin A, the transfer of vitamin A from pregnant mother to the fetus is carefully controlled. This results in all infants born with very low stores of vitamin A . Therefore human milk is still the best vitamin A source for infants. The concentration of vitamin A in breast milk is highest in the first 21 days postpartum (colostrum in the first 4-6 days and transitional milk in the next 7-21 days). Breast milk vitamin A concentrations and an infant's vitamin A status are based on maternal dietary intake. Breast milk retinol concentrations are a useful tool and a unique indicator for lactating women and represents extrapolations of vitamin A status of breastfed infant.

In high risk vitamin A deficiency areas, prior recommendation for lactating women was to give two doses of 200,000 IU vitamin A within 6 weeks post-delivery . However, the lack of impact evidence of this regimen led to the WHO's withdrawal of such recommendation as a public health policy .

Food-based intervention has been regarded as a sustainable approach to improve population vitamin A status. Most recently, vitamin A-depleted sows fed high-provitamin A carotenoid maize resulted in significant increase in liver stores in nursing piglets and significant higher milk retinol concentrations than sows fed white maize that given a high-dose vitamin A supplement .

Previous efforts to fortify staples or common vehicles with vitamin A offer promising solution to prevention of vitamin A deficiency in vulnerable population . Food fortified with vitamin A has potentials to improve women's vitamin A status and to increase the vitamin A concentrations of breast milk . Rice as the most important staple food in Thailand, represents the culture of consumption and lifestyle of Thai people . Recent study in Thai school children fed with extruded rice grains fortified with zinc, iron and vitamin A every weekday for 2 months, significantly increased liver stores of vitamin A, as assessed with a stable isotope technique . Likewise, fortification of rice with vitamin A may also benefit mothers during lactation.

The outcomes of this study will be useful to guide the promotion of food-based strategies to improve vitamin A status of mother and infant during lactation.

DETAILED DESCRIPTION:
Objectives To determine the efficacy of vitamin A fortified rice that gets into the breast milk of lactating mothers as determined by breast milk vitamin A concentrations, total body reserves of vitamin A via isotope dilution technique, following a 14 weeks feeding trial of lactating women.

Methodology The intervention will have two arms, vitamin A fortified rice and regular rice with 35 participants (lactating women) per group. Participants will receive one meal per day on weekdays for a period of 14 weeks. The fortified dose will be measured in the final cooked product, but we will aim to administer approximately 500 µg retinol in the rice meal. Vitamin A fortified rice is produced by extrusion technology by adding retinol into an artificial rice to be mix with the normal rice.

Data collection

1. Demographic data Each participants will be asked about demographic data in the first interview. The data includes general information (age, education and occupation), socioeconomic status, number of child and duration of breastfeeding mothers, if women had a child before.
2. Anthropometric data Anthropometric measurements include weight and height of participants and weight, length and head circumference of infants will be recorded in the first day and post-intervention.
3. Dietary assessment At the baseline (Day 1: 3+1 week after first breastfeed), all participants will be interviewed on food consumption in the previous 24 hours for 3 times (2 weekdays and 1 weekend day). The data consist of food items, food types, food components and weight or size of consumed portions. Information from the interviews will be analyzed by INMUCAL software (Mahidol University, Thailand)
4. Collection and analysis of breast milk sample Breast milk samples will be collected for vitamin A analysis. Collection of breast milk sample will be divided into two periods at the following time points which will start 3+1 week after first breastfeed.

   * at baseline: Day 1 and 15
   * 14 weeks post-intervention: Day 121 and 135
5. Collection and analysis of blood sample The change of vitamin A status of participants will be determined by using the pair13C-retinol isotope dilution test . This involves giving the first dose of 2 µmol retinol equivalent of 13C2-retinolretinyl acetate to participants on day 1 after that the second dose (2 µmol retinol) will be given to participants on the day 121. Blood sample will be collected 4 times (Day 1, 15, 121 and 135 after 3+1 week of first breastfeed) for measuring the isotopic ratio of 13C/12C and the calculation of liver vitamin A concentration. Blood samples will be drawn into plastic clot blood tubes and will be wrapped with aluminum foil for protection from light. Then, blood will be centrifuged at 3000 rpm for 15 minutes, serum will be separated immediately into dark cryovials and stored at -20 ◦c.

ELIGIBILITY:
Inclusion Criteria:

* free of diseases
* gestational age between 37 to 42 weeks
* willing to breastfeed for a period of 4-6 months

Exclusion Criteria:

* Hb > 70 g/L
* Postpartum Hemorrhage
* Twin, Baby with low birth weight
* Receiving vitamin A supplement during the study

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — lactation women
Enrollment: 70 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-24 (Estimated)

PRIMARY OUTCOMES:
Vitamin A liver store | 135 days
  vitamin A concentration per gram liver

SECONDARY OUTCOMES:
Breast milk retinol | 135 days
  vitamin A (retinol) concentration in breast milk
Serum retinol | 121 days
  Concentration of retinol in serum

OTHER OUTCOMES:
Hb | 135 days
  Hemoglobin concentration in whole blood
The gut microbiome | 135 days
  Changing of the composition of the microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Siwaporn Pinkaew, Ph.D, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Pattani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinkaew S, Udomkesmalee E, Davis CR, Tanumihardjo SA. Vitamin A-fortified rice increases total body vitamin A stores in lactating Thai women measured by retinol isotope dilution: a double-blind, randomized, controlled trial. Am J Clin Nutr. 2021 May 8;113(5):1372-1380. doi: 10.1093/ajcn/nqaa418. PMID 33675342